CLINICAL TRIAL: NCT06412705
Title: The Effect of Vit D on Post-extraction Site Bone Remodeling and Regeneration After 4 Months: A Prospective Clinical Trial
Brief Title: Vit D and Post-extractive Bone Turnover
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Studio Odontoiatrico Associato Dr. P. Cicchese e L. Canullo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VITD-01
Record Dates: First submitted 2024-05-05; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Vitamin D Deficiency; Alveolar Bone Loss; Alveolar Bone Resorption
Keywords: Dental Implants, Alveolar Bone Loss, Alveolar Process
MeSH Terms: conditions — Vitamin D Deficiency; Alveolar Bone Loss | interventions — Tooth Extraction; Dental Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tooth extraction and bone regeneration (Experimental): The present arm received tooth extraction and guided bone regeneration (performed with xenograft porcine material and collagen barrier membrane). After 4 months, a dental implant was inserted.
  Interventions: Procedure: Tooth extraction, guided bone regeneration and dental implant

INTERVENTIONS:
Procedure: Tooth extraction, guided bone regeneration and dental implant — The arm received tooth extraction and contextual guided bone regeneration. After 4 months, a dental implant was inserted.

SUMMARY:
The aims of the study was to correlate the extent of the dimensional alveolar bone changes after tooth extraction and contextual guided bone regeneration with serum vit D levels in 14 patients. Moreover, at 4 months, a small bone sample was collected in order to correlate histological and immunohistochemical parameters of bone with vit D serum levels.

DETAILED DESCRIPTION:
The study included 14 patients requiring tooth extraction and subsequent post-extraction bone regeneration with heterologous graft material of porcine origin. Four months after extraction, dental implants were placed, and insertion torque values (ITV) and implant stability quotients (ISQ) were recorded. During implant placement, a small bone sample was collected for histological analysis. The aim of the study was to analyze the correlation between serum vitamin D levels and post-extraction bone volume contraction, collagen type I (Col1A1), osteocalcin, osteopontin, runt-related transcription factor 2 (Runx2), ITV, ISQ, Newly Formed Bone Tissue (NFBT).

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult (≥ 18 years old)
* Patients willing to participate and to attend the planned follow-up visits

Exclusion Criteria:

* Absence of Type 1-Medical conditions requiring prolonged use of steroids and/or medications that can interfere with bone metabolism
* History of leukocyte dysfunction and deficiencies
* History of neoplastic disease requiring the use of radiation or chemotherapy
* History of renal failure
* Metabolic disorders such as osteoporosis and correlated vit D or antiresorptive medications assumption
* Physical handicaps that would interfere with the ability to perform adequate oral hygiene
* History of uncontrolled endocrine disorders
* Alcoholism or any drug abuse
* History of immunodeficiency syndromes
* Smoker of 10 cig per day, cigar equivalents or tobacco chewers
* Conditions or circumstances which in the opinion of the investigator would prevent completion of study participation or interfere with the analysis of the study results, such as history of non-compliance or unreliability
* Mucosa disease such as erosive lichen planus
* Residual post-extraction site with intact bone walls
* History of local irradiation therapy
* Persistent intraoral infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Dimensional alveolar bone changes | From extraction to implant insertion (4 months)
  Volumetrical changes of alveolar bone after tooth extraction measured by superimposition of two intraoral scans. The first was registered before the extraction of the tooth. The second was registered after 4 months (before inserting implant). The parameter used to measure the dimensional alveolar bone change is called "Integrated Distance" and it is expressed in mm3.
Evaluation of new formed bone tissue | Time of implant insertion: 4 months after extraction
  Evaluation of new formed bone tissue performed by histomorphometric methods.
Evaluation of Total Calcified Tissue (TCT) | Time of implant insertion: 4 months after extraction
  Evaluation of Total Calcified Tissue composed by the residual bone substitute utilized for regeneration plus the NFBT. The evaluation was performed by histomorphometrics methods.
Expression of Collagen A1 | Time of implant insertion: 4 months after extraction
  quantitative analysis of immunohistochemistry performed using deconvolution tool for ImageJ.
Expression of Osteocalcin | Time of implant insertion: 4 months after extraction
  quantitative analysis of immunohistochemistry performed using deconvolution tool for ImageJ.
Expression of Osteopontin | Time of implant insertion: 4 months after extraction
  quantitative analysis of immunohistochemistry performed using deconvolution tool for ImageJ.
Expression of Runx-2 | Time of implant insertion: 4 months after extraction
  quantitative analysis of immunohistochemistry performed using deconvolution tool for ImageJ.
Evaluation of Implant Stability Quotient (ISQ) | Time of implant insertion: 4 months after extraction
  Evaluation of Implant Stability Quotient after the implant insertion. The measurement was performed with "Osstell" system (W&H)
Evaluation of Implant Torque Value (ITV) | Time of implant insertion: 4 months after extraction
  Evaluation of Implant Torque Value at the implant insertion performed with the surgery implant device.

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Canullo, Principal Investigator — Studi Odontoiatrici Luigi Canullo
Locations (1):
- Studi Odontoiatrici Luigi Canullo, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No